CLINICAL TRIAL: NCT05166148
Title: Consequences of Eccentric Cycling on Exercise-related Neuromuscular Responses and Biomarkers in Breast Cancer Patients
Acronym: PROTECT-05
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-005
Record Dates: First submitted 2021-11-24; First posted 2021-12-21 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Eccentric Cycling; Physiological Responses
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- eccentric cycling compared to concentric cycling (Experimental): Every participant will perform the same protocol and will participated to the 3 experimental sessions (a, b and c) of the assigned intervention.
  Interventions: Other: Session (a); Other: Session (b); Other: Session (c)

INTERVENTIONS:
Other: Session (a) — Eccentric cycling
Other: Session (b) — High intensity concentric cycling realized at the same mechanical power output than eccentric cycling
Other: Session (c) — Low intensity concentric cycling realized at the same metabolic demand than eccentric cycling

SUMMARY:
This is a monocentric, prospective and interventional study aimed to investigating the physiological responses of eccentric compared to concentric cycling realized 1) at the same metabolic demand and 2) at the same mechanical power output. In order to compare the physiological responses between these two cycling modalities, 3 cycling sessions should be performed for each patient where concentric one will serve as reference / comparison to the eccentric one:

* Session (a): eccentric cycling
* Session (b): high intensity concentric cycling realized at the same mechanical power output than eccentric cycling
* Session (c): low intensity concentric cycling realized at the same metabolic demand than eccentric cycling The 3 sessions will be performed for each patient and order will be randomized.

DETAILED DESCRIPTION:
For each participant, 10 visits will be realized as followed:

Visit 1: determination of maximal O2 consumption (VO2max) and first familiarization session to eccentric cycling Visits 2, 3 and 4: second, third and fourth eccentric cycling familiarization sessions Visits 5, 7 and 9: cycling sessions (a), (b) and (c) attributed in a random order Visits 6, 8 and 10: post-24h measurements after cycling sessions

ELIGIBILITY:
Inclusion Criteria:

* Woman who completed (neo)adjuvant chemotherapy since less than 1 year for a breast cancer
* Woman under hormonotherapy, or menopausal woman, or woman in amenorrhea

Exclusion Criteria:

* Pregnant and nursing woman
* psychiatric, musculoskeletal or neurological disorders
* presenting at least one contraindication to the use of the transcranial magnetic stimulation
* presenting at least one contraindication to the realisation of the maximum effort test

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Investigate the physiological responses of the eccentric cycling on the knee extensors muscles by changes of neuromuscular parameters | 24 hours after pedaling sessions
  Measurement of neuromuscular fatigue via change in maximal voluntary isometric contraction of the knee extensors muscles registered via a force sensor.

SECONDARY OUTCOMES:
Comparison of muscle pain after eccentric in session (a) and after concentric modalities in session (b) and session (c) | 24 hours after pedaling sessions
  Measurement of muscle pain by visual analog scale (VAS) consists of a 100 mm long line providing a range of score from 0-100 (0: no pain, 100: worst possible pain).
Comparison of central (identified as a decrease in voluntary activation, VA) fatigue after eccentric in session (a) and after concentric modalities in session (b) and session (c) | 24 hours after pedaling sessions
  Measurement of central fatigue by percutaneous neurostimulation applied during the maximal voluntary contraction to evidence the level of voluntary activation (VA in %) and by transcranial magnetic stimulation to evidenced level of corticospinal excitability (measured by the MEP visible on EMG activity).
Comparison of peripheral (identified as a decrease in the quadriceps twitch muscle contractile capacities, Qtw) fatigue after eccentric in session (a) and after concentric modalities in session (b) and session (c) | 24 hours after pedaling sessions
  Measurement of peripheral fatigue by percutaneous neurostimulation applied at rest to evoked quadriceps twitch force (Qtw) to evidence muscle contractile properties.
Comparison of muscle thickness measured via ultrasonography on the vastus lateralis muscle after eccentric modality in pedaling session (a) and after concentric modalities in pedaling sessions (b) and (c) | 24 hours after pedaling sessions
  Change from baseline by ultrasonography measurements in the muscle thickness of the vastus lateralis muscle. Muscle thickness was measured as the distance from the superior border of the superficial aponeurosis and the superior border of the deep aponeurosis.
Comparison of muscle fibers pennation angle measured via ultrasonography on the vastus lateralis muscle after eccentric modality in pedaling session (a) and after concentric modalities in pedaling sessions (b) and (c) | 24 hours after pedaling sessions
  Change from baseline by ultrasonography measurements in the pennation angle of the vastus lateralis muscle. Pennation angle was measured as the angle between a fiber and the deep aponeurosis.
Comparison of muscle fibers fascile length measured via ultrasonography on the vastus lateralis muscle after eccentric modality in pedaling session (a) and after concentric modalities in pedaling sessions (b) and (c) | 24 hours after pedaling sessions
  Change from baseline by ultrasonography measurements in the fascicle length of the vastus lateralis muscle. Fascicle length was measured as the distance of a fibers between its insertion on the superficial aponeurosis and its insertions on the deep aponeurosis.
Comparison of muscle echogenecity measured via ultrasonography on the vastus lateralis muscle after eccentric modality in pedaling session (a) and after concentric modalities in pedaling sessions (b) and (c) | 24 hours after pedaling sessions
  Change from baseline by ultrasonography measurements in echogenecity of the vastus lateralis muscle. Echo intensity was determined based on the gray scale analysis of each pixel, the corresponding index of muscle quality ranging between 0 and 255 arbitrary units.
Comparison of blood markers in session (a) and after concentric modalities in session (b) and session (c) | 24 hours after pedaling sessions
  Change from baseline of blood markers dosage. Blood markers dosage investigated will: Reactive oxygen species (ROS), carbonylated protein, lipid peroxidation, antioxidant enzyme, proinflammatory cytokines, and muscle damage markers (creatine kinase, lactate dehydrogenase).

CONTACTS AND LOCATIONS:
Overall Officials: Roland SCHOTT, MD, Principal Investigator — Institut de cancérologie Strasbourg Europe
Locations (1):
- Institut de cancérologie Strasbourg Europe, Strasbourg, France